CLINICAL TRIAL: NCT01820598
Title: Acute and Medium-term Effects of Neuromuscular Electrical Multisite System (Kneehab®) on Cardiovascular Parameters and Induced Muscle Fatigue in Morbidly Obese Patients: Comparison With the Unidirectional Standard Device
Brief Title: Phase II Study of Neuromuscular Electrical Multisite System on Cardiovascular Effects in Severe Obese Patients
Acronym: StimobII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AGIR à Dom (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-AGIR-04
Record Dates: First submitted 2013-01-15; First posted 2013-03-29 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Arterial Stiffness; Electrical Stimulation; Training; Cardiovascular
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- m-NMES first (Other): Multisite electrostimulator first (Visit 1) and conventional electrostimulator then (Visit 2)
  Interventions: Device: Multisite NMES training during 6 weeks
- c-NMES first (Other): Conventional electrostimulator first (Visit 1) and multisite electrostimulator then (Visit 2)
  Interventions: Device: Multisite NMES training during 6 weeks

INTERVENTIONS:
Device: Multisite NMES training during 6 weeks
  Other Names: Kneehab(R) Stimulator

SUMMARY:
The study was designed to test the following hypotheses:

In patients with severe obesity, a multisite electrostimulation session (m-NMES) will induce higher changes in metabolic, inflammatory and cardiovascular parameters and higher increase in muscle strength during stimulated contractions than conventional unidirectional electrostimulation session (c-NMES).

In patients with severe obesity, a six-weeks m-NMES training program will enhance cardiovascular, metabolic and inflammatory parameters.

DETAILED DESCRIPTION:
Background: Physical activity is known to reduce cardiovascular risk as far as even minor change in lifestyle could occur. In obesity, physical activity programs remain challenging due to multifactorial causes related to body mass such as shortness of breath, traumatological pain or psychosocial causes. Although neuromuscular electrical stimulation training is presently ignored in the management of obesity, this technique may be appropriate and useful for muscle deconditioning in these patients. Furthermore, direct effects of electrostimulation training program on vascular function have been previously reported in spinal cord injury and chronic heart disease, suggesting that improvement in cardiovascular function may be expected. While a promising new technique of multisite electrical stimulation (the Kneehab® system) has been recently commercialized, few study have investigated the acute effects of electrostimulation on vascular function and not any study report the effects of electrical stimulation in obese patients.

MAIN OUTCOME OF THE ACUTE PHASE STUDY (1st part):To study the effect of multisite electrical stimulation session (m-NMES) on arterial stiffness as compared to conventional unidirectional electrical stimulation session (c-NMES) in patients with severe obesity. Secondary outcomes of the observational study: 1/ To study the effect of m-NMES on endothelial function, blood pressure, systemic inflammation and metabolic status (fasting glucose and insulin) as well as electrically-induced muscle fatigue as compared with c-NMES in patients with morbid obesity. 2/ To study the profile of responders to electrical stimulation according to body composition, 6-minute walking distance, spontaneous physical activity or susceptibility to tolerate electrical stimulation. Response to electrical stimulation will be assessed by an improvement in arterial stiffness after stimulation, if so.

MAIN OUTCOME OF THE INTERVENTIONAL STUDY (2nd part):To study the effect of a multisite electrical stimulation training program (m-NMES) (6 weeks, 30 sessions) on arterial stiffness in patients with severe obesity. Secondary outcomes of the interventional study: To study the effect of m-NMES on endothelial function, blood pressure, systemic inflammation and metabolic status (fasting glucose and insulin) as well as muscle strength, body composition, functional capacity (6-minute walking distance) and spontaneous physical activity, after 15 sessions (3 weeks) and after 30 sessions (6 weeks) of training program. Evaluation of the dose-response to m-NMES training in terms of arterial stiffness and functional capacity.

Expected outcomes: Acute change in arterial stiffness and/or endothelial function is expected after one m-NMES session and/or after c-NMES session. M-NMES session is expected to induce higher changes than c-NMES stimulation session on cardiovascular and muscle parameters. Chronic changes in arterial stiffness and/or endothelial function is expected after 6 weeks of m-NMES training.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 18 years
* Morbid obesity (BMI > 35 kg/m²)
* Not included into exercise training program in the year prior to inclusion- Spontaneous physical activity lower than 160 min wk (i.e. < 30 min/d x 5 d/wk).

Additional Inclusion criteria for the interventional study:

* Patients with PWV > 9.3 m / s

Exclusion Criteria:

* Underage- Pregnant or parturient women
* Persons deprived of their liberty for judicial or administrative reasons, person under a legal protection measure (article L1121-8)
* Exclusion period in other studies- Person not affiliated to a social security scheme
* Chronic alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Delta arterial stiffness | Day1 and Day3
  Change in carotid-femoral Pulse wave velocity (PWV) after NMES sessions

SECONDARY OUTCOMES:
Delta pulse arterial tonus (RH-PAT) | Day1 and Day3
  change in pulse arterial tonometry after NMES sessions
NMES-induced muscle fatigue | Day1 and Day3
  change in maximal voluntary contraction after NMES sessions
Delta blood pressure | Day1 and Day3
  changes in systolic and diastolic blood pressures after NMES sessions
Delta plasmatic biomarkers | Day1 and Day3
  changes in inflammatory and metabolic plasmatic biomarkers after NMES sessions
Body composition | Day1, Day21 and Day 42
  Fat-free mass and fat-free mass indexes assessed by impedancemetry
Spontaneous physical activity | Day1 and Day 42
  Number of hours per day of physical activity at 1, 2, 3, 4 or 5 metabolic equivalent(METS),Number of step per day,using a 7-days actigraphy
Maximal voluntary contraction | Day1, Day21 and Day 42
  Quadriceps peak force
Walking distance | Day1 and Day 42
  6-minute-walking test
Arterial stiffness | Day1, Day21 and Day 42
  Pulse wave velocity (PWV) measurements
Pulse artery tone (RH-PAT) | Day1, Day21 and Day 42
  Pulse artery tonometry measurement
Plasmatic biomarkers | Day1, Day21 and Day 42
  Inflammatory and metabolic biomarkers
Blood pressure | Day1, Day21 and Day 42
  Arterial systolic and diastolic blood pressure
Response to m-NMES | Day42
  Delta in current intensity during m-NMES between the first to the last session

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD, PhD, Principal Investigator — Laboratoire EFCR, CHU de Grenoble, 38043, Grenoble, France
Locations (1):
- Hopital Universitaire, Grenoble, France